CLINICAL TRIAL: NCT00474955
Title: Multicenter Open-label Observation Program in Patients With Chronic Hepatitis C and With Chronic Renal Failure (CRF) Receiving Peginterferon Alpha-2a (40 kDa) Pegasys
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Patients With Chronic Hepatitis C and Chronic Renal Failure.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20434
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- Peginterferon Alpha-2a (Experimental): Eligible participants will be administered peginterferon alpha-2a [Pegasys] (40 kilo Dalton), 180 micrograms as a subcutaneous injection, once in a week, for 48 weeks. Participants with a calculated glomerular filtration rate of <15 milliliter /minute will be administered a reduced dose of 135 mcg as a subcutaneous injection, once in a week, for 48 weeks.
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms or 135 micrograms sc weekly for 48 weeks

SUMMARY:
This single arm study will assess the efficacy and safety of PEGASYS in patients with chronic hepatitis C and end-stage renal disease, including patients on hemodialysis. Patients will receive PEGASYS at a dose of 180 micrograms weekly; those with a calculated glomerular filtration rate of <15mL/min will receive a reduced dose of 135 micrograms weekly. Following 48 weeks of treatment there will be a 24 week period of treatment-free follow-up. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-60 years of age;
* chronic hepatitis C;
* chronic renal failure, including patients on hemodialysis therapy;
* detectable HCV RNA levels (>500IU/mL).

Exclusion Criteria:

* concurrent active hepatitis A or B;
* history or evidence of a medical condition associated with chronic liver disease other than HCV;
* history or other evidence of decompensated liver disease;
* therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment <=6 months prior to study;
* acute renal failure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Russia (4):
  - Chita
  - Irkutsk
  - Khabarovsk
  - Orenburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 participants were enrolled in this study conducted from 2006 to 2011 at 5 centers in Russian Federation.
Groups:
- Peginterferon Alpha-2a: Eligible participants were administered peginterferon alpha-2a [Pegasys] [40 kilo Dalton (kDa)], 180 micrograms (mcg) as a subcutaneous injection, once in a week, for 48 weeks. Participants with a calculated glomerular filtration rate (GFR) of <15 milliliter (mL)/minute (min) were administered a reduced dose of 135 mcg as a subcutaneous injection, once in a week, for 48 weeks.
Period: Overall Study
Arm/Group | Peginterferon Alpha-2a
Started | 27
Completed | 19
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Drug unavailability | 1
Not completed — Personal reasons | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants who received at least one dose of study medication.
Groups:
- Peginterferon Alpha-2a: Eligible participants were administered peginterferon alpha-2a (40 kDa), 180 mcg as a subcutaneous injection, once in a week, for 48 weeks. Participants with a calculated GFR of <15 mL/min were administered a reduced dose of 135 mcg as a subcutaneous injection, once in a week, for 48 weeks.
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response at 24 Weeks Following Treatment Completion
Description: Sustained virologic response is defined as undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) levels (<50 international units [IU]/mL) at 24 weeks following the completion of 48 weeks treatment period (Week 72).
Time Frame: At Week 72
Population: ITT population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Percentage of participants | 55.6

2. Primary Outcome: Percentage of Participants With Undetectable Hepatitis C Virus Ribonucleic Acid Level at Week 24 and Week 48
Description: HCV RNA level less than 50 IU/mL was considered to be undetectable.
Time Frame: At Week 24 and Week 48
Population: ITT population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Percentage of participants
  At Week 24 | 59.3
  At Week 48 | 48.1

3. Primary Outcome: Percentage of Participants With At Least a 2log10 Drop in Hepatitis C Virus Ribonucleic Acid at Week 24 as Compared to Baseline
Description: The table below shows the percentage of participants with at least 2log10 drop in HCV RNA level at Week 24 as compared to Baseline (Screening visit [Days -30 to -1]).
Time Frame: From Baseline (Days -30 to -1) and Week 24
Population: ITT population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Percentage of participants | 33.3

4. Secondary Outcome: Number of Participants Who Experienced Any Adverse Events or Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect
Time Frame: Up to Week 72
Population: Safety population included all enrolled participants who received at least one dose of study medication, whether withdrawn prematurely or not, and who had at least one follow-up data point were included.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Participants
  Participants with any AEs | 10
  Participants with any SAEs | 2

5. Secondary Outcome: Number of Participants Who Prematurely Withdrew From the Treatment Over a Period of 48 Weeks
Description: Participants who prematurely withdrew from the treatment for the following reasons: personal reasons (not related to the study), adverse events, and drug unavailability, are presented.
Time Frame: Up to Week 48
Population: ITT population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Participants
  Personal reasons (not related to the study) | 5
  Adverse events | 2
  Drug unavailability | 1

6. Secondary Outcome: Number of Participants With Any Marked Abnormality in Laboratory Parameters Over a Period of 72 Weeks
Description: Marked abnormal laboratory parameters included serum glutamic pyruvic transaminase (SGPT), serum glutamic oxaloacetic transaminase (SGOT), gamma-glutamyl transpeptidase (GGTP), total bilirubin, alkaline phosphatase (ALP), ferritin and transferrin saturation. These laboratory parameters were evaluated at Baseline (Screening visit [Days -30 to -1]) and at various Visits (V): Week 0 (V1), Week 2 (V2), Week 4 (V3), Week 12 (V4), Week 24 (V5), Week 36 (V6) and Week 48 (V7) and after treatment completion at follow-up (FU) Week 4 (Week 52, V8), FU Week 12 (Week 60, V9), and FU Week 24 (Week 72, V10).
Time Frame: Up to Week 72
Population: ITT population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Participants
  SGPT Increased, Baseline | 6
  SGPT Increased, V1 | 5
  SGPT Increased, V2 | 4
  SGPT Increased, V3 | 4
  SGPT Increased, V4 | 6
  SGPT Increased, V5 | 8
  SGPT Increased, V6 | 5
  SGPT Increased, V7 | 2
  SGPT Increased, V8 | 4
  SGPT Increased, V9 | 3
  SGPT Increased, V10 | 3
  SGOT Increased, Baseline | 4
  SGOT Increased, V3 | 2
  GGTP Increased, V3 | 1
  Total bilirubin Increased, Baseline | 1
  ALP Increased Baseline | 7
  ALP Increased, V3 | 9
  Ferritin Increased, Baseline | 18
  Ferritin Decreased, Baseline | 1
  Ferritin Increased, V1 | 18
  Ferritin Increased, V4 | 17
  Ferritin Increased, V5 | 14
  Ferritin Increased, V7 | 14
  Transferrin saturation Increased, Baseline | 7
  Transferrin saturation Decreased, Baseline | 2
  Transferrin saturation Increased, V1 | 8
  Transferrin saturation Decreased, V1 | 1
  Transferrin saturation Increased, V4 | 7
  Transferrin saturation Increased, V5 | 4
  Transferrin saturation Decreased, V5 | 1
  Transferrin saturation Increased, V7 | 7

7. Secondary Outcome: Mean Change From Baseline in Blood Pressure up to Week 72
Description: Mean change from Baseline in diastolic blood pressure (DBP) and systolic blood pressure (SBP) was recorded at Baseline (Screening visit [Days -30 to -1]) and at various Visits (V): Week 2 (V2), Week 4 (V3), Week 12 (V4), Week 24 (V5), Week 36 (V6) and Week 48 (V7) and after treatment completion at follow-up (FU) Week 4 (Week 52, V8), FU Week 12 (Week 60, V9), and FU Week 24 (Week 72, V10).
Time Frame: From Baseline (Days -30 to -1) to Week 72
Population: ITT population included all enrolled participants who received at least one dose of study medication. Number of participants evaluable at a particular visit was determined by 'n'.
Measure: Mean (Standard Deviation); unit: Millimeter (mm) of Mercury
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Millimeter (mm) of Mercury
  DBP, V2, n=27 | -0.7 (8.6)
  DBP, V3, n=27 | 0.6 (12.1)
  DBP, V4, n=26 | -2.9 (7.2)
  DBP, V5, n=23 | -1.3 (10.1)
  DBP, V6, n=23 | -2.6 (9.0)
  DBP, V7, n=19 | -3.7 (9.6)
  DBP, V8, n=27 | -4.6 (8.1)
  DBP, V9, n=21 | -3.6 (9.1)
  DBP, V10, n=21 | -3.8 (9.2)
  SBP, V2, n=27 | -2.8 (12.9)
  SBP, V3, n=27 | 1.3 (15.6)
  SBP, V4, n=26 | -4.0 (11.6)
  SBP, V5, n=23 | -0.7 (12.0)
  SBP, V6, n=23 | -0.4 (10.3)
  SBP, V7, n=19 | -4.2 (13.2)
  SBP, V8, n=27 | -5.2 (11.3)
  SBP, V9, n=21 | -3.1 (17.4)
  SBP, V10, n=21 | -4.5 (14.7)

8. Secondary Outcome: Mean Change From Baseline in Heart Rate up to Week 72
Description: Mean change from baseline in heart rate was recorded at Baseline (Screening visit [Days -30 to -1]), and at various Visits (V): Week 2 (V2), Week 4 (V3), Week 12 (V4), Week 24 (V5), Week 36 (V6) and Week 48 (V7), and after treatment completion at follow-up (FU) Week 4 (Week 52, V8), FU Week 12 (Week 60, V9), and FU Week 24 (Week 72, V10).
Time Frame: From Baseline (Days -30 to -1) to Week 72
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Peginterferon Alpha-2a
Number analyzed (Participants) | 27
Beats per minute (bpm)
  V2, n=27 | 0.7 (4.9)
  V3, n=27 | 1.5 (4.2)
  V4, n=26 | 2.6 (7.9)
  V5, n=23 | 1.1 (5.6)
  V6, n=23 | 0.5 (6.0)
  V7, n=19 | 1.3 (6.4)
  V8, n=27 | 2.0 (5.2)
  V9, n=21 | 1.4 (3.1)
  V10, n=21 | -0.2 (4.4)

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: All SAEs and AEs were collected for safety population included all enrolled participants who received at least one dose of study medication, whether withdrawn prematurely or not, and who had at least one follow-up data point were included.
Arm/Group | Peginterferon Alpha-2a
Serious Adverse Events (participants affected / at risk) | 2/27
Other Adverse Events (participants affected / at risk) | 10/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alpha-2a (N=27)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Right acromioclavicular joint dislocation (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alpha-2a (N=27)
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Weber-Christian disease (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.